CLINICAL TRIAL: NCT04967976
Title: A Prospective Randomized and Controlled Study of Efficacy and Safety of TiLOOP® Bra Mesh in Patients With Expander-Implant Breast Reconstruction.
Brief Title: Breast Mesh Used in Two-staged Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E20210210
Record Dates: First submitted 2021-06-10; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Radiation; Breast Reconstruction; Synthetic Mesh
Keywords: breast cancer; breast reconstruction; radiation; synthetic mesh
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast Reconstruction with breast mesh (Experimental): The tissue expander-implant reconstruction with TiLoop Bra mesh.
  Interventions: Procedure: TiLoop Bra mesh in expander-implant breast reconstrution
- Breast Reconstruction without breast mesh (Active Comparator): The tissue expander-implant reconstruction without TiLoop Bra mesh. The tissue expander is placed sub-pectoral and covered by muscle/fascia.
  Interventions: Procedure: sub-pectoral expander-implant breast reconstruction

INTERVENTIONS:
Procedure: TiLoop Bra mesh in expander-implant breast reconstrution — The tissue expander is inserted with TiLoop Bra mesh in the first stage of reconstruction immediately after nipple/skin-sparing mastectomy. The tissue expander is placed sub-pectoral.
  Arms: Breast Reconstruction with breast mesh
Procedure: sub-pectoral expander-implant breast reconstruction — The tissue expander is inserted without TiLoop Bra mesh in the first stage of reconstruction immediately after nipple/skin-sparing mastectomy. The tissue expander is placed sub-pectoral and covered by muscle/fascia.
  Arms: Breast Reconstruction without breast mesh

SUMMARY:
This is the first prospective randomized and controlled study on the efficacy and safety of TiLOOP® Bra mesh in patients with expander-implant breast reconstruction. The investigators hypothesize that incoporating TiLOOP Bra mesh with tissue expanders will reduce the rates of capsular contraction, improve the efficiency of expansion and provide better aesthetic result.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with breast cancer
2. More than 18 years old
3. Karnofsky Performance Status (KPS) larger than 80
4. No clinical or imaging evidence of distant metastasis
5. BMI < 35kg/m2
6. Patients with no or mild breast ptosis
7. No severe deficiency in hematological, cardiovascular system, no immune-deficiency, no severe abnormal liver or kidney function.
8. Mental Health Patient

   -

   Exclusion Criteria:

1. Patients with distant metastasis of breast cancer or local recurrence; 2. Past ipsilateral breast/chest wall radiation; 3. Inflammatory breast cancer, stage IV breast cancer 4. History of severe allergic or specific constitution; 5. Mental illness; 6. Drug/alcohol abuse; 7. Pregnancy, lactation, or impregnated during the trial period; 8. Non-eligible to the study enrollment based on researchers' discretion

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Complication Rates | up to 24 months after surgery
  complications related to the reconstructed breast, including flap complications, capsular contracture, surgical site infection, prosthetic malposition/extrusion, reconstruction failure, etc.
Expansion Efficiency | through study completion, an average of 1 year
  percentage of average injected saline volume to total volume (E=average volume/ total volume）through study completion, an average of 1 year

SECONDARY OUTCOMES:
number of revision surgery | from the completion of expander exchange up to 24 months after surgery
  To record the rate of surgical revision events on the breast including but not limited to fat tranplantation, reduction mammoplasty/mastompexy, contralateral augmentation,
aesthetic outcome graded by Harris evaluation score and Breast-Q questionaire | from the completion of expander exchange up to 24 months after surgery
  Harris evaluation score was used to evaluate the aesthetic outcome of patients' reconstructed breasts, which was scored as "excellent," "good," "fair," "poor".
  Breast-Q questionaire was also used to evaluate the aesthetic outcome of patients' reconstructed breast.
psychological evaluation by Breast-Q questionnaire | from the completion of expander exchange up to 24 months after surgery
  We use the Breast-Q questionnaire to evaluate patients' satisfaction via the reconstruction module of BREAST-Q.
total cost | from expander implation up to the completion of expander exchange,through study completion, an average of 1 year
  total cost in RMB per captia
number of occurrence of deep venous thrombosis | from expander implation up to the completion of expander exchange, through study completion, an average of 1 year
  post-operative occurrence of deep venous thrombosis
number of occurrence of non-surgical site infection | from expander implation up to the completion of expander exchange, through study completion, an average of 1 year
  post-operative occurrence of non-surgical site infection including but not limited pneumonia, urinary tract infection, etc.

CONTACTS AND LOCATIONS:
Locations (6):
- MD Anderson Cancer Center, Houston, Texas, United States
- China (4):
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Jilin Cancer Hospital, Ch’ang-ch’un, Jilin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
- Technical University of Munich, Munich, Germany